CLINICAL TRIAL: NCT02487888
Title: Randomized, Blinded, Controlled Trial to EValuate the EcOnomic and ClinicaL Outcomes of Utilizing Genetic Testing to Improve Therapeutic Decision-Making COmpared to Empiric Prescribing as the StaNdard of Care
Brief Title: A Study of the Impact of Genetic Testing on Clinical Decision Making and Patient Care
Acronym: REVOLUTION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Proove Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PB008
Record Dates: First submitted 2015-06-26; First posted 2015-07-02 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Pain; Chronic Pain; Mental Disorders; Cardiovascular Diseases; Diabetes Mellitus, Type 2; Arthritis
Keywords: Genetic Variation; Genetic Polymorphism; Polymorphism, Single Nucleotide; Genetic Association Studies; Healthcare Utilization
MeSH Terms: conditions — Pain; Chronic Pain; Mental Disorders; Cardiovascular Diseases; Diabetes Mellitus, Type 2; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Pain (Experimental): Patients presenting to a clinic for pain, that will be either blinded to genetic testing results or unblinded to genetic testing results
  Interventions: Other: Unblinded to Genetic Testing Results; Other: Blinded to Genetic Testing Results
- Mental Health (Experimental): Patients presenting to a clinic for mental health disorders, that will be either blinded to genetic testing results or unblinded to genetic testing results
  Interventions: Other: Unblinded to Genetic Testing Results; Other: Blinded to Genetic Testing Results
- Cardiovascular (Experimental): Patients presenting to a clinic for cardiovascular complications, that will be either blinded to genetic testing results or unblinded to genetic testing results
  Interventions: Other: Unblinded to Genetic Testing Results; Other: Blinded to Genetic Testing Results
- Arthritis (Experimental): Patients presenting to a clinic for osteoarthritis or rheumatoid arthritis, that will be either blinded to genetic testing results or unblinded to genetic testing results
  Interventions: Other: Unblinded to Genetic Testing Results; Other: Blinded to Genetic Testing Results
- Type 2 Diabetes Mellitus (Experimental): Patients presenting to a clinic for T2DM, that will be either blinded to genetic testing results or unblinded to genetic testing results
  Interventions: Other: Unblinded to Genetic Testing Results; Other: Blinded to Genetic Testing Results

INTERVENTIONS:
Other: Unblinded to Genetic Testing Results — The physicians of this group of patients will be unblinded to the results of the genetic testing.
Other: Blinded to Genetic Testing Results — The physicians of this group of patients will be blinded to the results of the genetic testing. They will be un-blinded to the results of each patient once that patient has completed the study.

SUMMARY:
The purpose of this study is to evaluate the impact of genetic testing on healthcare decisions and patient outcomes for patients suffering from pain, cardiovascular problems, Arthritis, Type II Diabetes, and/or Mental Health disorders. Results of genetic testing will also be compared with the clinical outcome measures collected to discover novel genetic factors that may influence patient care.

DETAILED DESCRIPTION:
The molecular basis of many pharmacogenetic polymorphisms has now been elucidated, with genetic variations resulting in alteration of expression or function of receptors, enzymes, and transporters relevant to the safety and efficacy of a medical treatment. Genetics has been shown to be a significant factor in the variability of responses of medication choices and doses. With the rapid development of cost-effective high throughput molecular genotyping methods, pharmacogenetics has become increasingly important because of its potential to identify patients with increased risk of adverse drug reactions or decreased likelihood of response at standard dosage of drug. By identifying the genetic risks and the most effective therapy for an individual patient, clinicians may improve the efficacy of treatment and decrease the risk of adverse drug events. The addition of pharmacogenetic testing to routine clinical practice may also be extremely helpful because of the cost reduction associated with the identification of patients that will not respond to expensive drugs or with the identification of patients likely to suffer from severe adverse events. There are also tremendous efforts in the pharmaceutical industry to lower the cost for drug development; pharmacogenetics may fulfill the need to provide the right drug to the right patient and to increase the likelihood of success of large phase II and phase III clinical trials.

The purpose of this study is to evaluate how currently available genetic tests are being implemented in various clinics around the United States, and whether this information results in benefits to patient care. Patients presenting to clinics with pain, cardiovascular conditions, Arthritis, Type II Diabetes, and/or Mental Health disorders that are receiving Proove Bioscience's genetic testing will complete validated questionnaires to measure specific outcomes related to their treatment at each clinical visit, including medication efficacy, reduction in adverse drug events, and healthcare utilization. Physicians will document any changes made to treatment regimens, including adjustments to medications or non-pharmacological treatments, and any improvements in the outcome measures. Statistical analysis will be performed to calculate relationships between genotypic and phenotypic data points collected in this study.

The results of this study will provide a measurable understanding of the medical and economic value of implementing genetic testing into clinical care. Furthermore, data points collected will be used to examine novel correlations and associations between single nucleotide polymorphisms and longitudinal clinical outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or Female, at least 18 years of age
* Currently taking or a candidate for medication
* Documented or recent complaint within 90 days with initial date of onset

Exclusion Criteria:

* Severe hepatic or renal disease (where current pharmaceutical dosing is affected and/or requires adjustment of standard dosing prior to PGx testing)
* Significant diminished mental capacity that is unable to understand the protocol, surveys and questionnaires; unable to read/write English or Spanish.
* Recent febrile illness that precludes or delays participation by more than 1 month
* Pregnancy or lactation
* Participation in a clinical study that may interfere with participation in this study
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pain Scores on the Pain Numeric Rating Scale (NRS) | 60 days
Function/Disability assessment on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 60 days
Number of Participants that Experience of Adverse Events | Up to 2 years
Type of Adverse Events Experienced by Participants | Up to 2 years
Severity of Adverse Events Experienced by Participants | Up to 2 years
Type of medication or alternative therapy prescribed for participants, as listed on the Medication Efficacy Differentiation (MED) Scale or on the investigator's evaluation form | Up to 2 years
Medication dosage prescribed to the participants | Up to 2 years
Frequency of participant urine drug screens | Up to 2 years
Self-rated response levels to prescribed medications | 60 days
  Subjects are ask to rate the ability of their medication, on a scale of 0 to 5, to treat their condition and/or relieve their symptoms.
Presence and Severity of Generalized Anxiety Disorder on the GAD-2 | 60 days
Presence and Severity of Depression on the PHQ-2 | 60 days
Presence of atrial fibrillation symptoms and their impact on quality of life using the Severity of Atrial Fibrillation (SAF) scale | 60 days
Risk of cardiovascular incidents using the AHA Heart Disease Risk Assessment | 60 days
Risk of stroke using the CHA2DS2-VASc Score | 60 days
Severity of Rheumatoid Arthritis using the Routine Assessment of Patient Index Data (RAPID-3) score | 60 days
BMI for patients being treated for T2DM | 60 days
Glucose levels for patients being treated for T2DM | 60 days

SECONDARY OUTCOMES:
Co-occurring disorders collected by ICD-9/10 codes | 60 days
Assessment of previous treatments | 60 days
  Participants are asked to rate the benefit of previous treatments on a scale of 0 to 5.
Urine drug screen results | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Smith, M.D., Principal Investigator — G.S. Medical Center Inc./Comprehensive Pain Relief Group
Locations (31):
- United States (31):
  - Medical Clinic - Amy Weinberg M.D. Inc, Beverly Hills, California
  - Medical Clinic - Dr. Neil Ghodadra, Beverly Hills, California
  - Snibbe Orthopedics, Beverly Hills, California
  - Robert Graham, MD, Fresno, California
  - Bautista Medical Group, Fresno, California
  - Torrey Pines Orthopaedic Medical Group, La Jolla, California
  - Soha Dolatabadi Rheumatology, Los Angeles, California
  - Summit Family Medicine, Murrieta, California
  - Macer Medical, Rolling Hills, California
  - Medical Clinic - Paul C. Murphy, MD Inc, San Diego, California
  - Comprehensive Pain Relief Group, Torrance, California
  - The Doctor's Office, Vista, California
  - Medical Clinic - Dr. Kevin Monahan, MD, Boca Raton, Florida
  - Associates MD, Davie, Florida
  - Reeders Internal Medicine, Fort Lauderdale, Florida
  - Troutt & Associates, PSC, Fort Lauderdale, Florida
  - Medical Clinic - Kevin Ohayon MD Family Medicine, Fort Lauderdale, Florida
  - Neurology of Central Georgia, Macon, Georgia
  - Idaho Pain Clinic, Sandpoint, Idaho
  - Comprehensive Pain Clinic, Fort Wayne, Indiana
  - Medical Clinic - Dr. Rosenberg A. Reyes, Louisville, Kentucky
  - Interventional Pain Institute, Baltimore, Maryland
  - New England Center for Mental Health, Littleton, Massachusetts
  - Orthopedic Associates of SW Ohio, Vandalia, Ohio
  - Mallik Tella MD, Portland, Oregon
  - Lighthouse Medical, Altoona, Pennsylvania
  - Medical Clinic - Anthony Mathis, DPM, Greer, South Carolina
  - Personal Medicine, LLC, Chattanooga, Tennessee
  - Northgate Neurology, Hixson, Tennessee
  - Morristown Pain Consultants, Morristown, Tennessee
  - Pain Clinic of Spokane, Spokane, Washington